CLINICAL TRIAL: NCT00966758
Title: Open, Prospective Pilot Study to Obtain Aerosol Distribution in Asthmatic Patients Using SPECT-CT for Comparison With Functional Imaging Using Computer Methods
Brief Title: Open, Prospective Pilot Study to Obtain Aerosol Distribution in Asthmatic Patients Using Single Photon Emission Computed Tomography (SPECT) for Comparison With Functional Imaging Using Computer Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Prof Dr Wilfried De Backer, University Hospital Antwerp, Department of Respiratory Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PML_DOC_0901
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Computed Tomography; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Procedure: Computed Tomography — 1 low dose CT scan is taken
Procedure: Single Photon Emission Computed Tomography — 1 SPECT scan is taken

SUMMARY:
In this open prospective study, 6 well controlled asthmatic patients will undergo a high-resolution multi-slice computed tomography (CT) scan, lung function tests and a SPECT scan to obtain patient specific geometries of the central and peripheral small airways, patient specific boundary conditions and the in-vivo spatial distribution of inhaled aerosols.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with well controlled asthma as defined by the current GINA guidelines
2. Male or female patients aged ≥18 years
3. Patients with a documented positive response to the reversibility test (i.e. FEV1 increase ≥ 12% and 200mL from baseline value after 4 puffs of 100 µg of inhaled salbutamol pMDI) within the 12 months preceding the screening visit or performed at screening visit after a wash-out of 2 days for long acting β2 agonists or a documented positive response to the methacholine challenge test
4. Patients with a co-operative attitude
5. Written informed consent obtained
6. Patients maintained on stable respiratory medication for 4 weeks prior to visit 1

Exclusion Criteria:

1. Patients who are pregnant or are breast-feeding
2. Inability to carry out pulmonary function testing
3. Diagnosis of COPD as defined by the current GOLD guidelines
4. History of near fatal asthma
5. Hospitalization due to exacerbation or respiratory infection of the airways 4 weeks prior to visit 1
6. Current smokers or ex-smokers
7. Patients with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study
8. Cancer or any other chronic disease with poor prognosis and/or affecting patient status
9. BMI ≥ 35 kg/m2
10. Patients treated with CPAP or BiPAP
11. Known active tuberculosis
12. A history of cystic fibrosis, central bronchiectasis or interstitial lung disease
13. A history of thoracotomy with pulmonary resection
14. Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study
15. Patients who received any investigational new drug within the last 4 weeks prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Deposition of inhaled aerosol
  The primary objective of this study is to correlate the deposition distribution of inhaled aerosol obtained using computer methods through comparison with in-vivo SPECT data. The computer methods yield the concentration of particles entering and depositing in a lung lobe based on flow and particle behaviour simulation. The SPECT data yields the same parameter, i.e. particle concentration within each lung lobe, through scintigraphy assessment of the inhaled aerosols.

SECONDARY OUTCOMES:
Lobar aerosol deposition
  One of the secondary objectives is to assess the variability in lobar deposition between patients with both methods (CT and SPECT).
Sample size estimation for future studies
  Another secondary objective of this study is to establish a basis for a power calculation to determine adequate sample size for possible prospective studies.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried A De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium